CLINICAL TRIAL: NCT06783101
Title: A Pilot Randomized Controlled Trial: Utilizing a Digital Inhaler to Support Asthma Management in Adolescents With Intellectual and Developmental Disabilities
Brief Title: Using a Smart Inhaler to Support Asthma Management in Adolescents With Intellectual and Developmental Disabilities
Acronym: IDD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Responsible Party: Principal Investigator, Larry Yin, Associate Professor, Children's Hospital Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CHLA-24-00064
Record Dates: First submitted 2025-01-14; First posted 2025-01-20 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Asthma in Children; Intellectual Disabilities (F70-F79); Developmental Disability; Autism Spectrum Disorder (ASD)
Keywords: smart inhaler; asthma; inhaler proficiency; children; intellectual disability; developmental disability
MeSH Terms: conditions — Intellectual Disability; Developmental Disabilities; Autism Spectrum Disorder; Asthma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Standard asthma education arm
- Intervention (Experimental): Uses smart inhaler daily for 8 weeks
  Interventions: Behavioral: Use of smart inhaler to enhance asthma inhaler proficiency

INTERVENTIONS:
Behavioral: Use of smart inhaler to enhance asthma inhaler proficiency — The application of the smart inhaler technology to enhance asthma inhaler proficiency
  Arms: Intervention

SUMMARY:
Correct use of daily medications containing inhaled corticosteroids is key for asthma control, yet children with intellectual and developmental disabilities (IDD) face additional barriers to proper inhaler use. Smart inhalers, a novel technology that provides guidance and immediate feedback on inhaler use techniques, have been shown to enhance correct medication administration in the typically developing pediatric population, but their effectiveness has not been evaluated on the pediatric IDD population. This study aims to investigate whether daily application of smart inhalers (1) is feasible and acceptable in the IDD population, (2) improves the rate of correct medication administration, and (3) results in improvement in lung function. This effort aims to promote better asthma management in the IDD population.

DETAILED DESCRIPTION:
The study is a single-blinded randomized-controlled pilot trial with a goal of 30 participants ages 10-17 years diagnosed with IDD and moderate-to-severe asthma. Subjects are recruited from subspecialty clinics and a primary care FQHC at a large, urban academic children's hospital. Participants in the intervention group are assigned to use smart inhalers daily for 8 weeks, and the control group receives standard asthma education.

All participants attend three visits over 8 weeks, each scheduled four weeks apart. Primary outcomes, feasibility and acceptability, are assessed by data completeness and satisfaction surveys. Secondary outcomes, the Inhaler Proficiency Scales, are measured by the smart inhaler and by a trained observer and analyzed by Spearman's correlation test. Tertiary outcomes, Forced Expiratory Volume (FEV1) in one second, and Peak Expiratory Flow (PEF), are measured by a spirometer. Demographics and outcomes are reported as frequencies (%), mean (SD), or median (IQR). Analyses will utilize generalized linear mixed-effects models to account for the within-participant correlation.

ELIGIBILITY:
Inclusion Criteria: Participants must meet all of the inclusion criteria to participate in this study:

* Adolescents ages 10-17 years
* Diagnosis of mild-to-moderate intellectual disability: ICD-10: F70-F71 and/or diagnosis of developmental disability, including autism: ICD-10: F80-89
* Diagnosis of moderate-to-severe asthma or moderate or severe unspecified asthma: ICD-10: J45.40-J45.909
* Parent/legal guardian is willing to answer questions about their child.
* Parent/legal guardian and adolescent must have the ability to understand study procedures and to comply with them for the entire length of the study
* English or Spanish-speaking participants
* Not involved in other studies using digital inhalers
* Males and females of reproductive capability will be enrolled: contraception is not necessary or required.
* Participants must use any of the following MDIs (as indicated by the 510(k): Ventolin HFA, ProAir HFA, Advair HFA, Flovent HFA, Xopenex HFA, Symbicort HFA, Atrovent HFA, Proventil HFA, Alvesco HFA, Dulera HFA, and Asmanex HFA.

Exclusion Criteria: All candidates meeting any of the exclusion criteria at baseline will be excluded from study participation:

* Health status or any clinical conditions: Limited life expectancy, co-existing disease or other characteristics that precludes appropriate diagnosis, treatment, or follow-up in the trial.
* Inability or unwillingness of individual or legal guardian/representative to give written informed consent.

Ages: 10 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2024-08-13 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Feasibility of smart inhaler device | Weeks 1-8
  Feasibility will be determined by data completeness: Ratio of days on which there are valid smart inhaler data out of the total number of days
Acceptability of smart inhaler | Weeks 4 and 8
  Acceptability will be measured by response rate on user satisfaction survey.
Usability of smart inhaler | Weeks 4 and 8
  Usability will be measured by ease of use smart inhaler survey.

CONTACTS AND LOCATIONS:
Overall Officials: Larry Yin, MD, MSPH, Principal Investigator — Children's Hospital Los Angeles
Locations (1):
- Children's Hospital Los Angeles, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No